CLINICAL TRIAL: NCT00537524
Title: A Phase II, Randomized, Controlled, Observer-blind, Single-center Study to Evaluate the Immunogenicity, Safety and Tolerability of Two Doses of an H5N1 Influenza Vaccine in Subjects Aged 6 Months to 17 Years
Brief Title: Immunogenicity, Safety and Tolerability of Two Doses of a Pre-pandemic Influenza Vaccine in Participants Aged 6 Months to 17 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V87P6; 2007-002480-27
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Prophylaxis of Avian Influenza
Keywords: Bird flu; seasonal influenza vaccine; influenza vaccine; prepandemic vaccine; virus strain with the potential to cause pandemic; toddlers; children; adolescents
MeSH Terms: conditions — Influenza in Birds; Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): 0.5mL of H5N1 vaccine 7.5ug
  Interventions: Biological: H5N1 Influenza Vaccine
- Arm 2 (Active Comparator): 0.25 or 0.5mL of H5N1 vaccine
  Interventions: Biological: H5N1 Influenza Vaccine

INTERVENTIONS:
Biological: H5N1 Influenza Vaccine — Two 0.5mL injections of H5N1 influenza vaccine containing 7.5μg of H5N1 antigen (A/Vietnam/1194/2004), administered 3 weeks apart, and one 0.5mL injection of H5N1 vaccine 12 months after the second dose, IM into the deltoid muscle (preferably of the non-dominant arm) or anterolateral thigh (depending on the muscle mass).
  Arms: Arm 1
Biological: H5N1 Influenza Vaccine — Two 0.25mL or 0.5mL injections of H5N1 influenza vaccine, administered 3 weeks apart, IM into the deltoid muscle (preferably of the non-dominant arm) or anterolateral thigh (depending on the muscle mass).
  Arms: Arm 2

SUMMARY:
Evaluate the immune response and reactogenicity of H5N1 vaccination in subjects aged 6 months to 17 years compared to seasonal flu vaccination

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Receipt of Seasonal Influenza Vaccine for season 2007/2008
* Receipt of another vaccine within 3 weeks before and after each vaccination
* Previous vaccination with a pandemic candidate vaccine and/or vaccine containing the adjuvant MF59 or a similar adjuvant
* Children who are in the local recommendation for influenza vaccination due to underlying diseases

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 471 (Actual)
Dates: Start 2007-09; Primary Completion 2007-10 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of, and magnitude of antibody responses to two 0.5mL intramuscular injections of an H5N1 influenza vaccineapart | administered 3 weeks apart

SECONDARY OUTCOMES:
safety and tolerability of, and magnitude of antibodies to one booster dose with a H5N1 | 12 months after primary immunization
safety profile of a H5N1 compared to a seasonal flu vaccinepersistence of specific antibodies | 12 months after primary immunization

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- University of Tampere Medical School, Tampere, Finland

REFERENCES:
- [Result] Vesikari T, Karvonen A, Tilman S, Borkowski A, Montomoli E, Banzhoff A, Clemens R. Immunogenicity and safety of MF59-adjuvanted H5N1 influenza vaccine from infancy to adolescence. Pediatrics. 2010 Oct;126(4):e762-70. doi: 10.1542/peds.2009-2628. Epub 2010 Sep 6. PMID 20819892
- [Derived] Vesikari T, Forsten A, Borkowski A, Gaitatzis N, Banzhoff A, Clemens R. Homologous and heterologous antibody responses to a one-year booster dose of an MF59((R)) adjuvanted A/H5N1 pre-pandemic influenza vaccine in pediatric subjects. Hum Vaccin Immunother. 2012 Jul;8(7):921-8. doi: 10.4161/hv.20248. Epub 2012 Jul 1. PMID 22777094